CLINICAL TRIAL: NCT00570466
Title: Computer Based Intervention for Type 2 Diabetes in Youth: Phase 2
Brief Title: Computer Based Intervention for Type 2 Diabetes in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK66724 (completed); U44DK066724 (NIH); U01DK061231 (NIH)
Record Dates: First submitted 2007-12-06; First posted 2007-12-11 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2014-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Prevention; Children; Diet; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video games (Experimental): Two interactive, computer-based video games (9 sessions each) played in sequence to increase fruit, vegetable and water intake, physical activity and decrease TV viewing.
  Interventions: Behavioral: Video Games
- Web and DVD knowledge (Placebo Comparator): Parallel web and DVD based knowledge games on fruit, vegetable, water, physical activity and physical inactivity.
  Interventions: Behavioral: Web and DVD knowledge

INTERVENTIONS:
Behavioral: Video Games — Two interactive, computer-based video games (9 sessions each) played in sequence to increase fruit,vegetable,water intake + physical activity + decrease TV viewing.
  Arms: Video games
Behavioral: Web and DVD knowledge — Web and DVD based knowledge games
  Arms: Web and DVD knowledge

SUMMARY:
Interactive multimedia programs have been demonstrated to produce substantial change in children's dietary behaviors. This SBIR-Phase 2 protocol will evaluate the two video game interventions designed to change diabetes related behaviors, including diet and physical activity: Escape from Diab! and Nanoswarm that were developed in Phase 1. The primary hypotheses for this SBIR-Phase 2 protocol are:

1. The two video games will result in greater dietary and physical activity change than a knowledge based control group.
2. The effects of the video games will be mediated by changes in child preferences for FV and PA, self-efficacy to change FV intake and PA, and intrinsic motivation to eat FV and PA.

We will test these hypotheses by evaluating the two video games in a randomized experiment. To minimize costs, we will evaluate the impact of the games on behavior (diet and PA), BMI and related psychosocial variables, but not blood values. Our long-term goal is reducing the incidence of Type 2 diabetes and related health problems in youth.

DETAILED DESCRIPTION:
Increasing numbers of minority youth are at risk for developing Type 2 Diabetes (T2D) because of family history and overweight. While precise incidence and prevalence rates for T2D among children are not available, the prevalence has increased substantially in the last ten years, likely due to parallel increases in obesity among children. These cases are expected to progress to end organ damage at an early age, with the resultant increased personal and societal costs. Probable risk factors for T2DM include ethnicity (African American, Hispanic, Native American), family history of diabetes, and obesity. Prevention is key to reducing risks for T2D. The only modifiable risk factor is weight, which reflects dietary and physical activity practices. A diet high in fruit and vegetables, and appropriate in total calories and low in dietary fat are likely protective against both obesity and T2D. Although national data suggest the percentage of kilocalories (kcal) from fat consumed by children aged 2-17 decreased between 1989 and 1995 (now at 33% of total kcal), actual fat intakes did not decrease. Kcal intake, however, increased. Children's current intake of fruit and vegetables is less than one-half of the 5-A-Day goal. Changing the diet and physical activity practices to impact adiposity among children 10 to 12 years old before the onset of obesity or early in obesity holds great promise of preventing T2D. Furthermore, it is approximately this age that children assume more responsibility for their diet and physical activity, and thereby the intervention can be expected to have a greater impact on behavior. Children at the 50%tile or higher BMI are those most likely to progress to obesity, and thereby provide an important target group for obesity prevention.

Video games focused on promoting T2D-related changes in diet and physical activity, based on the most current theories of health behavior, hold the promise of preventing T2D among children, and thereby reducing lifelong disease burden. Unlike traditional media-based interventions (print, graphic, audio/visual, television broadcast), computer technology provides opportunities to influence behavior change through direct, personalized interactive experiences.

As part of a SBIR-Phase I, we created two video games: Escape from Diab! and Nanoswarm - Invasion from Inner Space. These intervention video games propose to increase fruit and vegetable intake to reduce total calories by displacing high fat, high calorie foods; increase water intake to decrease sweetened beverage consumption and total calories; increase physical activity; and decrease inactivity (e.g., TV watching, playing commercial video games). The behavioral and educational objectives address national behavior change objectives, including:

* Three to five servings of fruit (F) or 100% fruit juice (J) per day and Four to seven servings of vegetables (V) per day (based on child recommended calorie intake for age and weight),
* Five to eight glasses of water (W) per day,
* Moderate to vigorous Physical Activity (PA) of at least 60 min/day, and
* Physical Inactivity (PI) (TV, e-games, telephone) of no more than 2 hours per day.

Both games use an adventure storyline to capture the children's interest and attention, and thereby enhance their desire to keep coming back to the game across multiple sessions (between which behavior change goals are attempted). The storylines provide messages that reinforce the diet and physical activity change objectives. Seamlessly woven into each adventure session are programmed procedures for promoting behavior change (goal setting, goal review), which were tailored to characteristics of the child obtained through self report. Behavior change knowledge games, seamlessly woven into the storyline, are used to provide the basis for effective goal setting; and energy balance games, also seamlessly woven into the storyline, are used to provide the knowledge necessary to effectively self control caloric intake and output.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy 10-12 year old African-American, Hispanic-American, Anglo or Asian children.
2. Able to fluently speak, read and write English.
3. Able to play computer video games.
4. DSL or high-speed internet connection at home.
5. No dietary restrictions that limit their intake of fruit & vegetables or water.
6. No medical, physical handicaps or other reasons that would limit their physical activity.
7. Greater than 50% BMI, but less than 95% BMI.

Exclusion Criteria:

1. Children who are not in the target age range of 10-12 years old.
2. Not able to fluently speak, read and write English.
3. Not able to play computer video games.
4. No DSL or high-speed internet connection at home.
5. Dietary restrictions that limit their intake of fruit & vegetables or water.
6. Medical, physical handicaps or other reasons that would limit their physical activity.
7. Less than 50% BMI or greater than 95% BMI.
8. History of epileptic seizures.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dietary intake of servings of fruit and vegetables as measured by three 24-hour dietary recalls; and minutes of moderate to vigorous physical activity as measured by 5 days of accelerometry. | 6 months

SECONDARY OUTCOMES:
Height, weight, waist circumference, propylthiouracil (PROP) sensitivity status and nutrition and physical activity psychosocial questionnaires. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Baranowski, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Baranowski T, Baranowski J, Thompson D, Buday R, Jago R, Griffith MJ, Islam N, Nguyen N, Watson KB. Video game play, child diet, and physical activity behavior change a randomized clinical trial. Am J Prev Med. 2011 Jan;40(1):33-8. doi: 10.1016/j.amepre.2010.09.029. PMID 21146765